CLINICAL TRIAL: NCT06560307
Title: Examination of Programming with the Enterra® Therapy System in a Double-Blinded, Randomized, Prospective Study in the Treatment of Nausea and Vomiting Symptoms Using Gastric Electrical Stimulation
Brief Title: Study of Enhanced Programming Stimulation with the Enterra® Therapy System
Acronym: EXPEDITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enterra Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLN 001-PR-01218
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Gastroparesis; Gastroparesis Nondiabetic; Gastroparesis Due to Diabetes Mellitus
Keywords: Gastric electrical stimulation; Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Programming Stimulation (Active Comparator): Begin with nominal (lower stimulation) programming settings at Enterra Therapy System implantation. At treatment assignment, nominal programming will continue. Slight increases in device amplitude (stimulation) will be done at 3 Month visit and at later follow-up visits.
  Interventions: Device: Enterra Therapy System
- Enhanced Programming Stimulation (Experimental): Begin with nominal (lower stimulation) programming settings at Enterra Therapy System implantation. At treatment assignment, moderate increases in device amplitude (stimulation) and duty cycle (on/off cycles) will be done. Further adjustments to amplitude, duty cycle, and/or frequency (rate of pulses) will be done at follow-up visits.
  Interventions: Device: Enterra Therapy System

INTERVENTIONS:
Device: Enterra Therapy System — The Enterra® Therapy System for gastric electrical stimulation (GES) is indicated for the treatment of chronic intractable (drug refractory) nausea and vomiting secondary to gastroparesis of diabetic or idiopathic etiology in patients aged 18 to 70 years.
  Other Names: Gastric electrical stimulation

SUMMARY:
The purpose of this research study is to evaluate if an enhanced Enterra device programming strategy will improve symptoms associated with gastroparesis, improve symptoms in a faster amount of time, and improve quality of life measures.

Participants in this study will be evaluated for study entry criteria, have an Enterra Therapy System implanted, and be randomly assigned to one of two programming strategies. Participants will answer daily questions about their gastroparesis symptoms on an application with their phone/tablet. Participants will answer quality of life questionnaires about their gastroparesis symptoms at monthly study visits.

Participants will be involved in the study for up to six months after treatment assignment.

Programming parameters in the study are within currently approved labeling.

ELIGIBILITY:
Inclusion Criteria:

1. Completed informed consent process with signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged ≥18 or ≤70 years at time of Enterra® therapy implantation
4. Diagnosed with idiopathic or diabetic gastroparesis
5. Delayed solid-phase gastric emptying study (Eggbeaters™ test meal), completed within one year of patient enrollment in the study. Gastroparesis defined as > 60% retained at 2 hours and/or >10% retained at 4 hours
6. Investigator confirms normal endoscopy within one year of enrollment in the study
7. GCSI-DD score for nausea severity during the qualifying Baseline Period averaging 2.5 or more per week and vomiting averaging 5 or more episodes per week

Exclusion Criteria:

1. Post-surgical gastroparesis (e.g., fundoplication, Billroth I or II) or other active stomach or gastrointestinal diseases disorders which could explain symptoms in the opinion of the investigator
2. History of pyloroplasty or pyloromyotomy or G-POEM
3. Pregnancy or breastfeeding at the time of consent, or intent to become pregnant during the study
4. Active H. pylori infection
5. Significant hepatic injury (elevated ALT, AST, bilirubin)
6. Metabolic, mechanical, or mucosal inflammatory causes that may explain GI symptoms such as gallbladder disease, small bowel bacterial overgrowth, IBS, inflammatory bowel disease, celiac disease, liver or pancreatic disease, or bowel obstruction
7. Patients with significant cardiac or cardiovascular disease, malignancy, or other conditions
8. Participation in other clinical studies
9. Use of narcotics more than three days per week or other drugs that may affect motility (e.g., Glucagon-like peptide 1 (GLP-1) agonist drug)
10. Cannabis and/or cannabinoid use that exceeds either:

    1. Greater than 3 days of usage per week with 2 or less occurrences each day of use, or
    2. Greater than 3 grams of total usage per week
11. Previous diagnosis or history of orthostatic intolerance, e.g., POTS, neurocardiogenic syncope, orthostatic hypotension
12. Subject experiences discomfort during stimulation assessment that cannot be tolerated
13. Subjects with an underlying disease leading to follow-up by MRI outside of current MR conditional indications
14. Evidence of a failed response to temporary gastric electrical stimulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Vomiting Absolute Frequency | 3 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) weekly vomiting absolute frequency
Change in Nausea Severity Score | 3 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) nausea severity score

SECONDARY OUTCOMES:
Change in Vomiting Absolute Frequency | 6 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) weekly vomiting absolute frequency
Change in Nausea Severity Score | 6 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) nausea severity score
Change in Total Symptom Score | 3 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) total symptom score
Change in Total Symptom Score | 6 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) total symptom score
Change in Quality of Life Score | 3 Months
  As measured by the Patient Assessment of Upper Gastrointestinal Disorders Quality of Life (PAGI-QoL) score
Change in Quality of Life Score | 6 Months
  As measured by the Patient Assessment of Upper Gastrointestinal Disorders Quality of Life (PAGI-QoL) score
Change in Vomiting Absolute Frequency | 1 Month
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) weekly vomiting absolute frequency
Change in Nausea Severity Score | 1 Month
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) nausea severity score

CONTACTS AND LOCATIONS:
Overall Officials: Michael Awad, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (6):
  - University of South Florida, Tampa, Florida
  - University of Louisville, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Foundation for Surgical Innovation, Portland, Oregon
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No